CLINICAL TRIAL: NCT02861443
Title: Irrigation of the Large Intestine in the Patients With Colostomy : Epidemiology and Quality of Life
Acronym: IrriQOL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/MP-01
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-07

CONDITIONS: Colostomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: practice of colonic irrigation

SUMMARY:
The main objective of this study was to determine the frequency of the practice of colonic irrigation (CI) among patients with a colostomy,.

Other objectives are:

* To compare the quality of life between a group of patients with a colostomy and practicing CI versus a group of patients with a colostomy without CI.
* To determine the causes of non-realization of the CI or failure.
* To determine the conditions of realization of colonic irrigation by the return of user experience (time of day when the CI is practiced, amount and type of fluid used, time spent in the bathroom, time to recurrence of stool, media used between two irrigations).

ELIGIBILITY:
Inclusion Criteria:

* The subject was informed about the implementation of the study's objectives, constraints and the rights of the subject
* The subject is aged at least 18 years
* The subject is a member of the Ostomy Federation of France
* The subject has had a terminal colostomy for more than 6 months

Exclusion Criteria:

* The subject is under guardianship or curatorship
* The subject is under judicial protection
* The subject formalizes his/her opposition
* It is not possible to inform the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is composed of adults with end colostomy. The sample is drawn from adult members of "la Federation des stomisés de France" who have a terminal colostomy.
Sampling Method: Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Practice of large bowel irrigation (yes/no) | Day 0
  Does the patient practice large bowel irrigation? (yes/no)

REFERENCES:
- [Result] Boutry E, Bertrand MM, Ripoche J, Alonso S, Bastide S, Prudhomme M; French Federation of Ostomy. Quality of life in colostomy patients practicing colonic irrigation: An observational study. J Visc Surg. 2021 Feb;158(1):4-10. doi: 10.1016/j.jviscsurg.2020.07.003. Epub 2020 Aug 8. PMID 32782085